CLINICAL TRIAL: NCT06381934
Title: Validation of Diagnostic Indices to Simplify Hyponatremia Therapy Assessment - A Randomized, Controlled, Parallel-group Clinical Trial in Hospitalized Patients on Thiazide Diuretics (THAT Study)
Brief Title: Validation of New Diagnostic Indices to Simplify Hyponatremia Therapy Assessment in Patients on Thiazide Diuretics
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Basel, Switzerland (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2024-00335; kt23ChristCrain4
Record Dates: First submitted 2024-04-16; First posted 2024-04-24 (Actual); Last update posted 2026-02-11 (Actual); Status verified 2026-02

CONDITIONS: Thiazide Associated Hyponatremia
Keywords: Hyponatremia; Strong Apparent Ion Difference; Potassium Levels in Urine
MeSH Terms: conditions — Hyponatremia | interventions — Standard of Care

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Standard Care Group (Active Comparator): TAH patients randomised to the Standard Care Group will be followed by a physician not involved in the study.
  Interventions: Other: Standard Care
- aSID/ChU Guided Therapy Group (Active Comparator): TAH patients randomised to the aSID/ChU Guided Therapy Group will have aSID and ChU determined and, depending on the results, will be assigned to fluid administration with saline or drinking restriction.
  Interventions: Other: aSID/ChU Guided Therapy

INTERVENTIONS:
Other: Standard Care — Standard diagnosis and therapy procedures at physician's discretion.
  Arms: Standard Care Group
Other: aSID/ChU Guided Therapy — Stopping of thiazide therapy. Measure aSID:
  * aSID between 39 and 42 mmol/l : measure ChU
    * ChU lower than 15mmol/l : fluid administration (0.9% NaCl infusion, 250-500 ml over 2 hours followed by 10-20 ml/kg/24h)
    * ChU higher than 14.9 mmol/l : drinking restriction (of at least 50% of usual drinking volume)
  * aSID higher than 42 mmol/l : fuid administration (fluid administration (0.9% NaCl infusion, 250-500 ml over 2 hours followed by 10-20 ml/kg/24h)
  * aSID lower than 39 mmol/l : drinking restriction (of at least 50% of usual drinking volume)
  The aSID/ChU guided therapy will take place for a minimum of 1- and a maximum of 3 days after enrolment. Treatment and adherence to the treatment will be assessed and re-evaluated at least daily for 3 days or till discharge or sodium normalization.
  Arms: aSID/ChU Guided Therapy Group

SUMMARY:
This study is looking at two new parameters, aSID and ChU, to see if these can help physicians to distinguish between different causes of low sodium levels (hyponatremia) in Patients taking a medicament against high blood pressure (thiazide). Researchers also want to see if using these new parameters to decide on treatment works just as well, or better, than the current standard treatments.

DETAILED DESCRIPTION:
Thiazide or thiazide-like diuretics associated hyponatremia (thiazide associated hyponatremia, TAH) has a high prevalence in hospitalized patients. Patients might present either with a hypovolemic hyponatremia due to volume loss as a diuretic effect of thiazide, or with a syndrome of inadequate antidiuresis (SIAD) like hyponatremia in need of fluid restriction. Canonical urine indices are not useful in differential diagnosis, being directly influenced by thiazide itself. Current guidelines suggest the use of a clinical volume status assessment, but this approach has a poor diagnostic performance, with less than 50% of patients being rightly diagnosed thru that. The investigators showed in a retrospective analysis the possible role of strong apparent ion difference (aSID) and of chloride and potassium levels in urine (ChU) in differential diagnosis of TAH. The goal of this study is to investigate prospectively whether implementation of aSID and, in case of inconclusive aSID, ChU, allows a correct differential diagnosis and treatment of TAH.

ELIGIBILITY:
Inclusion Criteria:

* Hospitalized patients presenting at University Hospital Basel
* aged 18 years or older
* able to give informed consent as documented by signature
* with serum sodium level < 133 mmol/l and serum osmolality < 300 mOsm/kg
* with treatment with thiazide or thiazide-like diuretic

Exclusion Criteria:

* symptomatic hyponatremia in need of 3% hypertonic solution or intensive care treatment
* inability or contraindications to undergo the trial (i.e., any acute severe cardiovascular event requiring an immediate intervention)
* decompensated liver cirrhosis CHILD C
* decompensated heart failure NYHA III or higher
* severe valve impairment
* untreated adrenal insufficiency
* severe kidney disease in need of dialysis
* pregnancy or breastfeeding
* end of life care
* inability to follow the study procedures (i.e., language problem, dementia or critical illness).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 136 (Estimated)
Dates: Start 2024-05-06 (Actual); Primary Completion 2027-04 (Estimated); Study Completion 2027-04 (Estimated)

PRIMARY OUTCOMES:
Serum Sodium Level | at baseline, 24 hours and up to 72 hours
  Percentage of patients with an increase in serum sodium level > 4 mmol/l at day 1 or > 134 mmol/l in maximum 3 days in the aSID/ChU guided therapy group as compared to the standard care (control) group.

SECONDARY OUTCOMES:
Descriptive analyses: Changes in aSID in relation to changes in serum sodium levels | at baseline, 24 hours and up to 72 hours
  Descriptive analyses: Changes in aSID in relation to changes in serum sodium levels.
Descriptive analyses: Changes in ChU in relation to changes in serum sodium levels | at baseline, 24 hours and up to 72 hours
  Descriptive analyses: Changes in ChU in relation to changes in serum sodium levels.
Diagnostic performance analyses of: aSID and ChU | at baseline, 24 hours and up to 72 hours
  Sensibility, specificity, negative predictive value and positive predictive value at different cut-offs for adequate therapy of TAH. An adequate therapy of TAH is a therapy by which the patient reaches the primary endpoint independent from randomization arm.
Diagnostic performance analyses of: aSID measured in blood gas analysis | at baseline, 24 hours and up to 72 hours
  Sensibility, specificity, negative predictive value and positive predictive value at different cut-offs for adequate therapy of TAH. An adequate therapy of TAH is a therapy by which the patient reaches the primary endpoint independent from randomization arm.
Diagnostic performance analyses of: clinical volume status assessment | at baseline, 24 hours and up to 72 hours
  Sensibility, specificity, negative predictive value and positive predictive value at different cut-offs for adequate therapy of TAH. An adequate therapy of TAH is a therapy by which the patient reaches the primary endpoint independent from randomization arm.
Diagnostic performance analyses of: not-invasive instrumental volume status assessment | at baseline, 24 hours and up to 72 hours
  Sensibility, specificity, negative predictive value and positive predictive value at different cut-offs for adequate therapy of TAH. An adequate therapy of TAH is a therapy by which the patient reaches the primary endpoint independent from randomization arm.
Diagnostic performance analyses of: other hormones such as aldosterone, renin, arginine-vasopressin | at baseline, 24 hours and up to 72 hours
  Sensibility, specificity, negative predictive value and positive predictive value at different cut-offs for adequate therapy of TAH. An adequate therapy of TAH is a therapy by which the patient reaches the primary endpoint independent from randomization arm.

CONTACTS AND LOCATIONS:
Overall Officials: Laura Potasso, Dr. med. sc., Principal Investigator — University Hospital, Basel, Switzerland
Locations (1):
- University Hospital Basel, Basel, Switzerland

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Vogt K, Widmer D, Kirsch M, Christ-Crain M, Potasso L. Validation of new diagnostic indices to simplify hyponatremia therapy assessment in patients on thiazide diuretics: study protocol of a randomized, controlled, parallel-group trial (THAT-Study). Trials. 2025 Jul 11;26(1):242. doi: 10.1186/s13063-025-08925-4. PMID 40646556